CLINICAL TRIAL: NCT02951858
Title: Screening and Brief Interventions for Substance Use in Primary Medical Institution
Brief Title: Substance Use Screening Among Drug User
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, DU, Jiang, Cheif Physician, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JDu-003
Record Dates: First submitted 2016-10-23; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Substance Use
Keywords: Alcohol,Smoking,and Substance Use Involvement Screening Test; Brief Intervention; Substance Use; Primary Medical and Health Care Institution
MeSH Terms: conditions — Substance-Related Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): The medical staffs who received the training will use the manual of brief intervention to deliver it and other materials about the harm of substance use.
  Interventions: Behavioral: Intervention Group
- Control Group (Active Comparator): The participants only receive the materials about the harm of substance use.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Intervention Group — The medical staffs who received the training will use the manual of brief intervention to deliver BI and other materials about the harm of substance use.
  Arms: Intervention Group
Behavioral: Control Group — The participants only receive the materials about the harm of substance use.
  Arms: Control Group

SUMMARY:
The purpose of this research is to improve the ability of primary medical staffs in screening and intervention for alcohol, benzodiazepines, and other illicit drug use.

DETAILED DESCRIPTION:
In order to reduce the social and personal harm caused by drugs, it is urgent to strengthen the ability of the primary health institutions in screening and intervention the addictive substances use. Firstly, the investigators will invite 10 primary medical staffs and 10 experts in addition to revise the manual of Alcohol, Smoking, and Substance Use Involvement Screening Test (ASSIST) and Brief Intervention (BI). Then, the investigators will recruit 100 medical staffs to participate the training of ASSIST and BI. Secondly, the researcher will investigate the effects of BI technology in reducing the use of addictive substances, improve the addiction related knowledge of patients through randomized controlled study. Finally, the investigators will collect the research information, revise the manual, and promote the training.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-60 years;
2. the patient to the community medical institutions;
3. ASSIST score is in 12-27, in a moderate risk;
4. voluntary to participate;
5. to agree to complete baseline interviews and follow-up studies.

Exclusion Criteria:

1. unable to complete the questionnaire;
2. serious physical illness, action inconvenience.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Risk Behaviors measured by ASSIST questionnaire | 1 month
  Risk Behaviors will be measured by ASSIST questionnaire.
Knowledge related to Substance Use measured by Knowledge related to Addiction questionnaire | 1 month
  Knowledge related to substance use will be measured by Knowledge related to Addiction questionnaire.
Motivation measured by Pre-treatment Readiness Scale | 1 month
  Motivation will be measured by Pre-treatment Readiness Scale (PRS).

SECONDARY OUTCOMES:
Depression measured by Self-Rating Depression Scale | 1 month
  the change of depression will be measured by Self-Rating Depression Scale (SDS).
Anxiety measured by Self-Rating Anxiety Scale | 1 month
  the change of anxiety will be measured by Self-Rating Anxiety Scale (SAS).
Self-esteem measured by Self-esteem questionnaire | 1 month
  the change of self-esteem will be measured by Self-esteem questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Du, M.D, Principal Investigator — Shanghai Mental Health Center

IPD SHARING:
Plan to Share IPD: No